Statistical Analysis Plan

Investigating the Effectiveness of an Entertainment Education Short Film for Internalized HIV

Stigma Reduction, Intimate Partner Status Disclosure Intentions, and Antiretroviral Medical

Adherence Intentions: A Randomized Controlled Trial Among Black Women Living with HIV

in the Southern U.S.

ClinicalTrials.Gov Identifier: NCT03898063

February 15, 2021

## **Introduction: Purpose of the Statistical Analysis Plan (SAP)**

The purpose of this Statistical Analysis Plan (SAP) is to detail the study objectives, study hypotheses and research questions, as well as the primary outcome measures and data analyses.

## **Study Overview**

This randomized controlled trial was conducted among Black women living with HIV in the Southern U.S. between the ages of 18 and 50. The study examined the efficacy of a short entertainment education (EE) narrative in comparison to a standard brochure for primarily improving the following: HIV status disclosure intentions, internalized HIV-related stigma, and antiretroviral medical adherence. Once consented, all participants completed a pre-test survey. Upon completing the pre-test, using the randomization feature in Qualtrics, participants were randomly assigned to one of two study arms: 1) EE narrative or 2) Brochure. After viewing the EE stimulus or the brochure, participants immediately completed a post-test survey. The primary aim of the study is listed below.

**Aim 1**. To investigate the effectiveness of an EE intervention for decreasing internalized HIV-stigma and increasing HIV status disclosure intentions and medical adherence intentions among Black women living with HIV in the Southern U.S.

The hypotheses guiding this research study included the following:

H<sub>1a-c</sub>: Participants in the EE condition will report: a) lower levels of internalized stigma; b) higher levels of disclosure intentions; c) higher levels of medical adherence intentions.

## **Data Collection Plan**

Participants will be recruited via two primary methods. Firstly, Facebook advertisements will be deployed to recruit participants who meet the inclusion criteria. Secondly, participants will be recruited via a Qualtrics panel.

## **Statistical Methods**

An Analysis of Covariance (ANCOVA) will be used to control for the influence of age on the relationships of interest. This analysis will determine if there is a statistically significant difference between the treatment arm (90 DAYS film) and the control arm (Brochure) on the following primary variables: internalized stigma, intentions to disclose, and intentions for medical adherence. The analyses will be conducted using SPSS version 24.